CLINICAL TRIAL: NCT04447391
Title: Effects of a 12-week Combined Exercise Program on Acylated and Desacyl Ghrelin, and Ghrelin O Acyl Transferase in Obese Adolescent Girls
Brief Title: Effects of a 12-week Combined Exercise Program on Ghrelins in Obese Adolescent Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 04-2015-015
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Ghrelin

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Exercise group who performed a combined exercise and 300 kcal/day deficit diet during 12 weeks.
  Interventions: Other: Combined exercise program
- Control group (Placebo Comparator): Control group who performed 300 kcal/day deficit diet during 12 weeks.
  Interventions: Other: Control

INTERVENTIONS:
Other: Combined exercise program — Combined exercise programme, consisting of warm-up, aerobic exercise, resistance training, and cool-down, 3 days a week after school for 50 minutes from 17;30 under supervision by a trainer plus 300 kcal deficit diet
  Arms: Exercise group
Other: Control — 300 kcal deficit diet only
  Arms: Control group

SUMMARY:
This study aimed to explore the effects of a 12-week combined exercise on ghrelin O acyl transferase, acylated ghrelin and desacylated ghrelin levels in obese girls.

DETAILED DESCRIPTION:
Little is known about on ghrelin O acyl transferase (GOAT), acylated ghrelin (AG) and desacylated ghrelin (DAG) levels during long-term exercise in adolescent population. Our previous study showed that combined exercise program in overweight children increases DAG with unchanged AG. This study aimed to explore the effects of a 12-week combined exercise on GOAT, AG, and DAG in obese girls.

ELIGIBILITY:
Inclusion Criteria:

* girls between 16 and 18 years
* being classified as being overweight or obese defined with the 85th percentile of body mass index or above based on the 2007 growth chart for Korean children aged 2-18 years.
* After consultation with a physician, they were required to be considered physically healthy enough to engage in regular exercise after school.

Exclusion Criteria:

* participation in any weight-management programme in the past 6 months
* engagement in other exercise programs except for regular physical education at school
* smoking
* amenorrhea for consecutive 2 months or more
* being treated for hereditary diseases, mental disorder, hypertension, diabetes mellitus, or musculoskeletal impairments
* taking any medication or supplements for weight control

Ages: 16 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09-10 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
body fat percent | Change from baseline body fat percent at 12 weeks
  Changes in body fat percent during 12 weeks
acylated ghrelin | Change from concentrations of baseline acylated ghrelin at 12 weeks
  Changes in concentrations of acylated ghrelin during 12 weeks
desacylated ghrelin | Change from concentrations of baseline desacylated ghrelin at 12 weeks
  Changes in concentrations of desacylated ghrelin during 12 weeks

SECONDARY OUTCOMES:
ghrelin O acyl transferase | Change from baseline concentrations of ghrelin O acyl transferase at 12 weeks
  Changes in concentrations of ghrelin O acyl transferase during 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeungsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No